CLINICAL TRIAL: NCT06844487
Title: Phase 3, Randomised Maternal and Infant (From 4 to 24 Months of Age) Safety and Immunogenicity Trial of MVA-BN® Vaccine in the Democratic Republic of the Congo
Brief Title: Phase 3 Infant Safety & Immunogenicity Trial of MVA-BN® in DRC
Acronym: PregInPoxVac
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jean-Pierre Van geertruyden (Other)
Collaborators: Ace Africa (Other); PENTA Foundation (Network); Bavarian Nordic (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of Kinshasa (Other); CEPI (Other)
Responsible Party: Sponsor-Investigator, Jean-Pierre Van geertruyden, Prof. Dr, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PIPVac-001 Infant Component
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-02

CONDITIONS: Mpox (Monkeypox); Vaccination; Immunogenicity; Safety; Infants; Children
Keywords: MVA-BN; Monkeypox virus; mpox; Infants; Children; Non-inferiority testing; Paediatric; Phase 3; Vaccine; Smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; Randomised
MeSH Terms: conditions — Mpox, Monkeypox; Smallpox

STUDY DESIGN:
Intervention Model Description: 344 male or female infants/children will be randomised (1:1) to receive the two doses of the standard MVA-BN vaccine, administered 28 days apart (N= 172), or two half doses of the standard MVA-BN vaccine, administered 28 days apart (N= 172).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child group 1 (Active Comparator): Male or Female infants/children aged 4-24 months will be administered each vaccine of the MVA-BN standard or half-dose regimen (depending on the randomisation group) by SC administration into the anterolateral thigh. For children closer to 24 months old, the deltoid of the upper arm can also be used (preferably the nondominant arm, if already known).
  Interventions: Biological: MVA-BN standard regimen
- Child group 2 (Active Comparator): Male of female infants/children aged 4-24 months will be administered each vaccine of the MVA-BN standard or half-dose regimen (depending on the randomisation group) by SC administration into the anterolateral thigh. For children closer to 24 months old, the deltoid of the upper arm can also be used (preferably the nondominant arm, if already known).
  Interventions: Biological: MVA-BN half-dose regimen
- Historical arm (Other): Historical data from healthy adults aged 18 to 50 years old, and children aged 2 to <12 years old from the POX-MVA-045 study (NCT06549530), will be used for safety and immunogenicity comparisons. These participants will be vaccinated in the deltoid of the upper arm.
  Interventions: Biological: MVA-BN standard regimen

INTERVENTIONS:
Biological: MVA-BN standard regimen — The MVA-BN vaccine, with the active ingredient: Modified Vaccinia Ankara-Bavarian Nordic, will be administered as a standard two-dose regimen at 1x10^8 TCID50 Inf.U./0.5 mL. The doses will be given 28 days apart (±3 days) via subcutaneous injection into the deltoid muscle, preferably in the non-dominant arm.
  Arms: Child group 1; Historical arm
Biological: MVA-BN half-dose regimen — The MVA-BN vaccine, with the active ingredient: Modified Vaccinia Ankara-Bavarian Nordic, will be administered as two half doses of the standard regimen; meaning infants/children allocated to Child Group 2 will receive 0.25 mL of the 0.5 mL. 1x10^8 TCID50 Inf.U./0.5 mL standard regimen. The doses will be given 28 days apart (±3 days) via subcutaneous injection into the deltoid muscle, preferably in the non-dominant arm. Only one vial will be used per infant/child.
  Arms: Child group 2

SUMMARY:
This Phase 3 double-blinded, randomized study aims to evaluate the safety and immunogenicity of the two-dose MVA-BN mpox vaccine regimen, administered subcutaneously, in infants and children aged 4 to 24 months in the Democratic Republic of the Congo (DRC), a population at high risk of mpox infection and complications. The study will compare the safety and immunogenicity of a full-dose regimen versus a half-dose regimen in this population. A hierarchical testing strategy will be applied as follows: first, non-inferiority of the full-dose regimen in infants/children (4-24 months old) will be evaluated against the full-dose regimen in adults from the POX-MVA-045 study. If non-inferiority is demonstrated, the immunogenicity of the half dose in infants/children (4-24 months old) will subsequently be tested for non-inferiority vs the full dose in adult. The trial will be conducted in Boende, Tshuapa Province, DRC.

The trial plans to enroll 344 male and female infants/children, who will be randomized to receive two doses of the MVA-BN vaccine administered 28 days apart. Participants in Child Group 1 (N=172) will receive the standard vaccine dose (0.5 mL), while those in Child Group 2 (N=172) will receive half the standard dose (0.25 mL), with both groups following the same dosing schedule.

This study builds on positive safety and immunogenicity data from prior trials that support the use of the standard dose regimen in younger children. However, considering the developmental differences in the immune systems of infants and young children/adolescents, it aims to evaluate whether a half-dose regimen can provide similar immunogenicity while potentially reducing reactogenicity. The findings will offer valuable insights into the optimal dosing strategy for this age group, balancing safety and immunogenicity to inform future vaccination recommendations.

DETAILED DESCRIPTION:
This Phase 3 double-blinded, randomised study aims to evaluate the safety and immunogenicity of the MVA-BN mpox vaccine regimen, administered subcutaneously, in infants and children aged 4 to 24 months in the Democratic Republic of the Congo (DRC), a population at high risk of mpox infection. The study will compare the safety and immunogenicity of a full-dose regimen versus a half-dose regimen. A hierarchical testing strategy will be applied as follows: first, non-inferiority of the full-dose regimen in infants/children (4-24 months old) will be evaluated against the full-dose regimen in adults from the POX-MVA-045 study. If non-inferiority is demonstrated, the immunogenicity of the half dose in infants/children (4-24 months old) will subsequently be tested for non-inferiority vs the full dose in adult.

The study will be conducted at the General Reference Hospital of Boende, Tshuapa Province, DRC.

The trial plans to enroll 344 male and female infants/children, who will be randomized to receive two doses of the MVA-BN vaccine administered 28 days apart. Participants in Child Group 1 (N=172) will receive the standard dose of the MVA-BN vaccine (1x10⁸ TCID50 Inf.U./0.5mL), while those in Child Group 2 (N=172) will receive half the standard dose (0.5x10⁸ TCID50 Inf.U./0.5mL). Participants randomized to receive the full dose will receive 0.5 mL of the MVA-BN vaccine, while participants randomized to receive the half dose will receive 0.25 mL of the MVA-BN vaccine.

During the screening visit, parents or legal guardians of the infant/child will provide informed consent and must pass a test of understanding (TOU) to confirm eligibility, with up to three attempts permitted. Demographics, medical history, and vaccination history will be recorded. A basic physical examination will be performed to assess general appearance, key organ systems, growth measurements (weight, length, and head circumference), neurological reflexes, and behavior. Vital signs (heart rate, respiratory rate, temperature, and blood pressure) will also be measured, and an HIV test will be performed.

Randomization will occur after eligibility is confirmed. Participants will be assigned to one of two groups through a double-blind randomization design. A block randomization method will ensure balanced allocation between the two groups, with randomization lists securely provided to unblinded personnel responsible for vaccine preparation. Blinding procedures will ensure that neither parents/legal guardians nor reactogenicity investigators know the group assignments.

Whenever possible, the first vaccine dose (Day 0) will be administered on the same day as the screening visit. However, vaccination may be postponed if the child has a fever or acute infection.

On Day 0, participants will undergo a physical examination, and their vital signs and vaccination/medication history will be assessed. A malaria test will be performed. Blood samples will be collected for baseline immunogenicity testing, including neutralizing antibodies, total binding antibodies, and IgG-binding antibodies.

Participants will then receive their first vaccine dose, administered subcutaneously (standard or half dose, based on randomization). Parents/legal guardians will be provided with a participant journal to document solicited AEs (e.g., pain, swelling, redness at the injection site, fever, irritability) and unsolicited AEs.

On day seven (Day 7), the Parents/legal guardians will be asked to return with the participant journal to report the data on (un)solicited AEs collected during the week after the first dose. Ongoing AEs will continue to be followed until resolution.

On Day 28, participants will undergo a physical examination, and their vital signs, vaccination history, and medication history will be reviewed, and malaria test will be performed. Parents/legal guardians will be asked about unsolicited AEs since the first vaccination. If no concerns are identified, participants will receive the second vaccine dose, and a new participant journal will be provided to document any AEs.

On Day 35, the Parents/legal guardians will be asked to return with the participant journal to report the data on (un)solicited AEs collected during the week after the second dose. Ongoing AEs will continue to be followed until resolution.

On Day 42, Participants will have a physical examination, including assessments of growth, developmental milestones, and general health. Blood samples will be collected to assess neutralising antibodies and total binding antibodies.

Day 56 any unsolicited AEs occurring between Day 35 and Day 56 will be followed up via telephone call or home visit.

On Day 208 (6 months after the second dose), Participants will return for a follow-up assessments, including a physical examination and evaluations of growth and developmental milestones. Vaccination and medication history will also be reviewed. Blood samples will be collected to assess long-term immune responses, including neutralizing antibodies and (total) binding antibodies.

On Day 395 (one year after the second dose), the final follow-up visit will focus on a comprehensive physical examination of the infant/child. Blood samples will be collected to assess long-term immune responses, including neutralizing antibodies and (total) binding antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be between 4 and 24 months old upon enrolment.
2. The participant's parent or legal guardian must pass (≥9/10) the TOU after being advised of the risks and benefits of the trial in a language understood by the parent/guardian and before performing any trial-specific procedures.

   - Note: If the participant's parent or guardian fails the TOU test on the first attempt, he/she must be retrained on the purpose of the study and must take the test again (2 repeats are allowed). If the participant's parent/guardian fails on the third attempt, the screening or consenting procedures should not continue.
3. The participant's parent or guardian must sign and date the informed consent form after reading the form and being advised of the risks and benefits of the trial in a language understood by the participant and before performing any trial-specific procedures.
4. The participant must live in the Boende health zone or its surrounding health zones in the Tshuapa province of the DRC.
5. The participant must be generally healthy in the investigator's clinical judgment and on the basis of vital signs assessed at day 1 screening with no severe (chronic) conditions (as far as medically known) that might interfere with vaccine assessment.

   - Note: HIV-positive subjects can be enrolled as long as their general condition is good, i.e., they are on antiretroviral treatment or have no signs or symptoms of immunosuppression, diagnosed on the basis of physical examination, medical history, and the investigator's clinical judgment.
6. The participant's parent(s) or guardian(s) of the child must agree to follow the study protocol, including attending follow-up visits and reporting any adverse events.
7. The participant must be available and his/her parent(s) or guardian(s) must be willing to have their child participate for the duration of the study.

The participant's parent(s) or guardian(s) must be willing to provide verifiable identification and have means to be contacted (phone number or address).

Exclusion Criteria:

1. The child is excluded if their mother received the MVA-BN vaccine during her pregnancy with the child or during the immediate postpartum period while breastfeeding the child.
2. Known history of cowpox, mpox or vaccinia infection.
3. Close contact in the 2 weeks prior to signing the ICF with anyone known to have mpox.
4. Known history of or active autoimmune disease (vitiligo or thyroid disease requiring thyroid replacement are not exclusions), history of Guillain-Barré syndrome or Reye's syndrome.
5. Having received any smallpox or licensed or investigational poxvirus-based (e.g. ACAM2000, MVA-BN based like MVA-BN-Filo) vaccine in the past.
6. Must not have received another experimental or non-licensed vaccine within 4 weeks before receiving the MVA-BN vaccine and during the trial.
7. Known allergy or history of anaphylaxis or other severe adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg, egg products and aminoglycosides.
8. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., tris(hydroxymethyl)-amino methane, including a history of allergic asthma.
9. Acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of responses, including but not limited to neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions.

   - Note: Participants with minor acute illnesses such as mild diarrhoea or mild upper respiratory tract infection or temperature ≥38.0ºC at screening will be excluded from enrolment at that time but may be rescheduled for re-screening later if feasible.
10. Presence of significant medical conditions or clinically significant findings at screening or vital signs for which, in the opinion of the gynaecologist, participation would not be in the best interest of the participant (e.g., compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments.

    * Note: Participants who have recently received treatment for acute, uncomplicated malaria are eligible for participation if at least 3 days have elapsed from the conclusion of a standard, recommended course of therapy for malaria; participants who are acutely ill with malaria at the time of screening should complete therapy and wait an additional 3 days after completion before screening for the study.
    * Note: Participants with sickle cell trait can be included.
11. History of malignancy (e.g., leukaemia, lymphoma).
12. Chronic administration (defined as more than 14 days) of systemic high dose immune-suppressant drugs (2 mg/kg/day or more of prednisolone or its equivalent or 20 mg/day or more for children who weigh more than 10 kg) from 6 months prior to first trial vaccination to trial conclusion.

    - Note: Participants receiving antiretroviral (ARV) medication for the management of HIV infection are eligible for inclusion, provided they meet inclusion criterion 5.
13. Major surgery (per the investigator's judgment) within the 4 weeks before screening or planned major surgery during the study (from the start of screening onwards).
14. Post-organ and/or stem cell transplant, whether or not with chronic immunosuppressive therapy.
15. Administration or planned administration of immunoglobulins and/or any blood products from 3 months prior to the first trial vaccination until the visit at the end of the active trial period (packed red blood cells given for an emergency indication in an otherwise healthy person and not required as ongoing treatment is not exclusionary [e.g., packed red blood cells given in an emergency during elective surgery]).
16. Received an investigational or nonregistered drug or vaccine or used an invasive investigational or nonregistered medical device within 30 days prior to vaccination or current or planned participation in another clinical study during the study.

    - Note: Participation in an observational clinical study is allowed.
17. History of chronic urticaria (recurrent hives).
18. The parent/legal guardian has employment with the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or relationship to the investigator or study site employee.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 344 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of Full-Dose vs. Half-Dose MVA-BN Vaccine in Infants/Children. | 14 days after the second dose
  Compare the immunogenicity of full-dose and half-dose MVA-BN vaccine regimens in infants/children (4-24 months), with neutralising antibody responses measured by PRNT assays 14 days post-second dose, against the full-dose regimen in adults from the POX-MVA-045 study.
  A hierarchical testing strategy will be applied as follows: first, non-inferiority of the full-dose regimen in infants/children (4-24 months old) will be evaluated against the full-dose regimen in adults from the POX-MVA-045 study. If non-inferiority is demonstrated, the immunogenicity of the half dose in infants/children (4-24 months old) will subsequently be tested for non-inferiority vs the full dose in adult.
Safety and Reactogenicity of the MVA-BN Vaccine in Infants/Children Compared to Adults from the POX-MVA-045 Study | Throughout the trial period; from the first dose to one year after the second dose
  Evaluate the safety and reactogenicity of the standard MVA-BN regimen administered subcutaneously to infants/children (4-24 months), compared to the standard regimen in adults from the POX-MVA-045 study. Safety endpoints include SAE, AESI, MAAE, and AE occurrences; reactogenicity endpoints include solicited local and systemic events.

SECONDARY OUTCOMES:
Immunogenicity of Standard and Half-Dose Regimens in Infants/Children vs. Adults and Older Children. | From baseline to one year after the second dose
  To assess the immunogenicity of the MVA-BN standard and half dose regimen administered subcutaneously (SC) in eliciting neutralising antibodies in infants/children (4-24 months old) compared to adults and children (2-<12 years old) of the POX-MVA-045 study receiving the standard MVA-BN regimen at baseline and all collected timepoints after the second dose.
Total Binding Antibody Response in Infants/Children vaccinated with MVA-BN Vaccine standard regimen and adults and children of the POX-MVA-045 study | From baseline to one year after the second dose
  To assess the immunogenicity of the MVA-BN standard and half dose regimen administered subcutaneously (SC) in eliciting total binding antibodies in infants/children (4-24 months old) compared to adults and children (2-<12 years old) of the POX-MVA-045 study at baseline and all collected timepoints after the second dose.
Immunogenicity of Standard vs. Half-Dose Regimens in Infants/Children. | From baseline to one year after the second dose
  To assess the immunogenicity of the MVA-BN standard versus half dose regimen administered subcutaneously (SC) in eliciting neutralising antibodies in infants/children (4-24 months old) at baseline and all collected timepoints after the second dose.
Total Binding Antibody Response with Standard vs. Half-Dose Regimens in Infants/Children. | From baseline to one year after the second dose
  To assess the immunogenicity of the MVA-BN standard versus half dose regimen administered subcutaneously (SC) in eliciting total binding antibodies in infants/children (4-24 months old) at baseline and all collected timepoints after the second dose.
Safety and Reactogenicity of Standard vs. Half-Dose MVA-BN Vaccine in Infants/Children. | Throughout the trial period; from the first dose to one year after second dose
  To evaluate the reactogenicity and safety of the MVA-BN standard regimen administered SC to infants/children (4-24 months old) compared to infants/children (4-24 months old) receiving the half dose regimen.
Safety and Reactogenicity of Standard MVA-BN Vaccine in Infants/Children Compared to Older Children. | Throughout the trial period; from first dose to one year after second dose
  To evaluate the reactogenicity and safety of the MVA-BN standard regimen administered SC to infants/children (4-24 months old) compared to children 2 to <12 years-old receiving the standard regimen (POX-MVA-045).

OTHER OUTCOMES:
Impact of Demographic Variables on Neutralising Antibody Responses in Infants/ Children Vaccinated with Half-Dose Regimen | From enrolment to one year after the second dose
  To explore demographic variables (e.g. age, sex, malaria exposure, malnutrition, etc.) that impact the neutralising and total binding antibody response in the serum of infants/children (4-24 months old) vaccinated with the half-dose MVA-BN regimen.
Impact of Demographic Variables on Total Binding Antibody Responses with Standard Regimen | From enrolment to one year after the second dose
  To explore demographic variables (e.g. age, sex, malaria exposure, malnutrition, etc.) that impact of neutralising and total binding antibody response against vaccinia in the serum of infants/children (4-24 months old) vaccinated with the standard MVA-BN regimen.
Neutralising Antibody Response in Standard and Half-Dose Regimens in a Subset of Infants/Children. | From baseline to one year after the second dose
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the monkeypox and vaccinia virus in a subset (10%) of 4 to 24-month-old infants/children compared to a subset (10%) of infants/children receiving a half-dose regimen (0.5 x108 TCID50 Inf.U./0.5mL) at baseline, 2 weeks, 6 months and 12 months after the second dose.
Total IgG Response Against Multiple MPXV Antigens with Standard and Half-Dose Regimens. | From enrolment to 1 year after the second dose
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting Total IgG in serum with multiple MPXV specific antigens (B6R, B2R, E8L, M1R, A35, H3L) in a subset (10%) of 4 to 24-month-old infants/children compared to a subset (10%) of infants/children receiving a half-dose regimen (0.5 x108 TCID50 Inf.U./0.5mL) at baseline, 2 weeks, 6 months and 12 months after the second dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Boende Hôpital Général de Référence, Boende, Boende, La Tshuapa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemey G, Lariviere Y, Zola TM, Maketa V, Matangila J, Mitashi P, Vermeiren P, Thys S, De Bie J, Muhindo HM, Ravinetto R, Van Damme P, Van Geertruyden JP. Algorithm for the support of non-related (serious) adverse events in an Ebola vaccine trial in the Democratic Republic of the Congo. BMJ Glob Health. 2021 Jun;6(6):e005726. doi: 10.1136/bmjgh-2021-005726. PMID 34183329
- [Background] Zola Matuvanga T, Lariviere Y, Lemey G, De Bie J, Milolo S, Meta R, Esanga E, Vermeiren PP, Thys S, Van Geertruyden JP, Van Damme P, Maketa V, Matangila J, Mitashi P, Muhindo-Mavoko H. Setting-up an Ebola vaccine trial in a remote area of the Democratic Republic of the Congo: Challenges, mitigations, and lessons learned. Vaccine. 2022 May 31;40(25):3470-3480. doi: 10.1016/j.vaccine.2022.04.094. Epub 2022 May 9. PMID 35550847
- [Background] Puri A, Pollard AJ, Schmidt-Mutter C, Laine F, PrayGod G, Kibuuka H, Barry H, Nicolas JF, Lelievre JD, Sirima SB, Kamala B, Manno D, Watson-Jones D, Gaddah A, Keshinro B, Luhn K, Robinson C, Douoguih M; EBL4001 Study Group. Long-Term Clinical Safety of the Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: A Prospective, Multi-Country, Observational Study. Vaccines (Basel). 2024 Feb 17;12(2):210. doi: 10.3390/vaccines12020210. PMID 38400193
- [Background] Lariviere Y, Zola T, Stoppie E, Maketa V, Matangila J, Mitashi P, De Bie J, Muhindo-Mavoko H, Van Geertruyden JP, Van Damme P. Open-label, randomised, clinical trial to evaluate the immunogenicity and safety of a prophylactic vaccination of healthcare providers by administration of a heterologous vaccine regimen against Ebola in the Democratic Republic of the Congo: the study protocol. BMJ Open. 2021 Sep 28;11(9):e046835. doi: 10.1136/bmjopen-2020-046835. PMID 34588237
- [Background] Poland GA, Kennedy RB, Tosh PK. Prevention of monkeypox with vaccines: a rapid review. Lancet Infect Dis. 2022 Dec;22(12):e349-e358. doi: 10.1016/S1473-3099(22)00574-6. Epub 2022 Sep 15. PMID 36116460
- [Background] Beeson AM, Haston J, McCormick DW, Reynolds M, Chatham-Stephens K, McCollum AM, Godfred-Cato S. Mpox in Children and Adolescents: Epidemiology, Clinical Features, Diagnosis, and Management. Pediatrics. 2023 Feb 1;151(2):e2022060179. doi: 10.1542/peds.2022-060179. PMID 36471498
- [Background] Sanchez Clemente N, Coles C, Paixao ES, Brickley EB, Whittaker E, Alfven T, Rulisa S, Agudelo Higuita N, Torpiano P, Agravat P, Thorley EV, Drysdale SB, Le Doare K, Muyembe Tamfum JJ. Paediatric, maternal, and congenital mpox: a systematic review and meta-analysis. Lancet Glob Health. 2024 Apr;12(4):e572-e588. doi: 10.1016/S2214-109X(23)00607-1. Epub 2024 Feb 21. PMID 38401556
- [Background] Bunge EM, Hoet B, Chen L, Lienert F, Weidenthaler H, Baer LR, Steffen R. The changing epidemiology of human monkeypox-A potential threat? A systematic review. PLoS Negl Trop Dis. 2022 Feb 11;16(2):e0010141. doi: 10.1371/journal.pntd.0010141. eCollection 2022 Feb. PMID 35148313
- See also: MVA-BN — https://www.bavarian-nordic.com/pipeline/technology/mva-bn.aspx
- See also: MVA-BN Product Characteristics — https://www.ema.europa.eu/en/documents/product-information/imvanex-epar-product-information_en.pdf